CLINICAL TRIAL: NCT01485471
Title: Spectroscopic Evaluation of Middle Ear Infection
Brief Title: Spectroscopic Evaluation of Middle Ear Infection (Withdrawn)
Status: Withdrawn | Type: Observational
Why Stopped: No paticipants enrolled
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Elliot Botvinick, Ph.D., Assistant Professor, Biomedical Engineering, University of California, Irvine
Other Study IDs: 20108015
Record Dates: First submitted 2011-08-02; First posted 2011-12-05 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Middle Ear Infection
Keywords: Middle Ear Infection
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medical Tool: Diffuse optical spectroscopy imaging ear exam
  Interventions: Device: Diffuse optical spectroscopy imaging

INTERVENTIONS:
Device: Diffuse optical spectroscopy imaging — ear exam imaging

SUMMARY:
Otitis media is more common in young children and it is estimated that 75% of all children experience at least one episode before the age of three. Otitis media is one of the common pediatric diagnoses and recurrent episodes account for the most commonly performed surgical procedure. Despite this a high degree of inaccuracy exists in diagnosis of this condition which depends on subjective assessment of the ear drum via direct visualization using an otoscope. Researcher can use Diffuse optical spectroscopy and diffuse optical imaging for the analysis of ear drum and the middle ear.

DETAILED DESCRIPTION:
The research can use low energy laser signal light from Diffuse optical spectroscopy that is harmless to the tissues and sends them into the ear canal to measure the tissue optical properties including the absorption of the laser signal and the amount of signal that will be backscattered by the ear drum. These measurements will then be analyzed using a microprocessor to determine presence of fluid or inflammation of the eardrum.

Diffuse optical spectroscopy an imaging method use near- infrared light to measure absolute tissue concentrations of oxyhemoglobin, deoxyhemoglobin, water, and lipids, as well as subtle changes in water and protein binding states

ELIGIBILITY:
Inclusion Criteria:

1. Male/ female at all age- newborn to adult.
2. Non- pregnant woman.
3. Diagnose of middle ear infection and plan for surgery procedure.

Exclusion Criteria:

1. Pregnant woman
2. Incompetent adults (i.e. individuals with cognitive impairment)
3. No diagnose of middle ear infection and no plan for surgery procedure.
4. Adults with cognitive impairment and children of parents that are cognitively impaired and thus are unable to consent will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UCI otolaryngology clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Middle Ear exam | 6 hours
  Diffuse optical spectroscopy imaging to evaluate ear drum

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Botvinick, Ph.D, Principal Investigator — Beckman Laser Institute; Bruce Tromberg, PhD, Study Director — Beckman Laser Institute